CLINICAL TRIAL: NCT02330653
Title: A Phase I/II, Double Blinded, Placebo Controlled, Single-center Study of Fecal Microbiota Transplant (FMT) for the Treatment of Active Pediatric Ulcerative Colitis and Pediatric Active Crohn's Colitis
Brief Title: Fecal Microbiota Transplant (FMT) in Pediatric Active Ulcerative Colitis and Pediatric Active Crohn's Colitis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Stacy A. Kahn (Other)
Responsible Party: Sponsor-Investigator, Stacy A. Kahn, Associate Director of the Inflammatory Bowel Disease Center, Boston Children's Hospital
Organization: Boston Children's Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P00014876; NCT02330211 (obsolete NCT alias)
Record Dates: First submitted 2014-12-29; First posted 2015-01-05 (Estimated); Results first posted 2023-10-16 (Actual); Last update posted 2023-10-16 (Actual); Status verified 2023-10

CONDITIONS: Inflammatory Bowel Diseases; Ulcerative Colitis; Crohn Disease
Keywords: Colitis; Fecal Microbiota Transplant; Ulcerative colitis; inflammatory bowel disease; Crohn's Disease
MeSH Terms: conditions — Inflammatory Bowel Diseases; Colitis, Ulcerative; Crohn Disease; Colitis | interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Fecal Microbiota Transplant (FMT) (Experimental): Induction retention enema for the first week of treatment followed by once weekly administration of 15 capsules of study treatment (the equivalent of 7.5 grams of human stool) will be (administered within 60 minutes of thawing once weekly) for 7 weeks. After completing 8 weeks of blinded study treatment, study subjects on FMT who have shown improvement will be given the option to receive open-label maintenance FMT weekly for an additional 8 weeks of once weekly FMT capsule administration.
  Interventions: Biological: Fecal Microbiota Transplant (FMT)
- Placebo (Placebo Comparator): Induction placebo enema for the first week of treatment followed by once weekly administration of 15 capsules of study placebo (administered within 60 minutes of thawing once weekly) for 7 weeks. After completing 8 weeks of blinded study placebo, study subjects on placebo who DO NOT demonstrate improvement will be given the option to receive open-label maintenance FMT weekly for an additional 8 weeks, beginning with a FMT induction enema followed by 7 weeks of weekly FMT capsule administration.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Fecal Microbiota Transplant (FMT) — The study intervention consists of frozen, bottled or encapsulated fecal microbiota preparations that have been screened and prepared to a uniform and rigorous standard by OpenBiome. FMT is performed by patients receiving a retention enema and swallowing capsules, introducing stool from a healthy donor into their intestinal tract.
  Other Names: Screened, healthy human donor stool
  Arms: Fecal Microbiota Transplant (FMT)
Biological: Placebo — Placebo administration will consist of both a placebo retention enema and placebo capsules.
  Arms: Placebo

SUMMARY:
The primary aims of this phase I/II, randomized, placebo controlled study are the assessment of safety and tolerability of universal donor FMT compared to placebo in pediatric and young adult subjects (ages 5 years through 30 years) with active ulcerative colitis (UC) or active Crohn's colitis (CD) who have failed, are intolerant to, or have refused traditional first-line maintenance therapy. Secondary objectives include the identification biomarkers in both donor and recipient that may confer a clinical response and to establish whether or not ongoing FMT maintenance therapy is required for maintenance of clinical benefit in pediatric UC or pediatric CD.

DETAILED DESCRIPTION:
This is a single-center pilot, phase I/II, randomized, prospective, double-blinded, placebo-controlled study of FMT in the treatment of active pediatric UC and active pediatric CD. The primary aim is to assess safety and feasibility of a weekly FMT maintenance therapy. A total of 10 patients with active UC (as defined by PUCAI score of >9) and 10 patients with active CD (as defined by PDCAI score of >10) will be enrolled and randomized to receive FMT or placebo-FMT (study treatment) by retention enema for 1 week and oral, frozen encapsulated inocula/placebo for 7 weeks. After the first 8 weeks, subjects on FMT who improve or subjects on placebo-FMT who do not improve will have the option to continue on study treatment or switch to open-label FMT until the end of 4 months from study initiation. Subjects will be followed by telephone to assess adverse events for a total of 6 months after their last FMT dose.

An initial subset of no more than 20 subjects will be enrolled in the study (will be limited to only those patients 12 years of age or older and to those who have mild to moderate disease) and randomized to receive FMT or placebo. We'd expect short term adverse events to occur within 7 days of FMT administration. Individual subject safety data will be reviewed by the PI to assess whether FMT appears to be safe in the subject before continuing the subject towards open-label use of FMT.

Patient metadata and stool samples will be collected at key time points. The patient-reported metadata collection technique will allow for numerous clinical correlations to be parsed out using the random forest machine learning capabilities of synthetic learning in microbial ecology (SLiME) to identify taxonomic features associated with important clinical parameters.

ELIGIBILITY:
Male and female children and young adults, aged 5 years to 30 years, who meet the following inclusion criteria, will be enrolled in the study.

Two initial subsets will be created: an initial subset of 20 subjects limited to patients greater than or equal to 12 years of age with mild to moderate ulcerative colitis (i.e., PUCAI < 65) patients with mild to moderate Crohn's disease (i.e., PDCAI less than or equal to 30).

All patients must satisfy below criteria:

1. Have UC (PUCAI >9) or CD (PDCAI >10) and have failed, are intolerant to, or have refused first-line maintenance therapy.
2. Have had visual or histologic evidence of inflammation confirmed through colonoscopy no more than 105 days prior to randomization.
3. Have negative test results for Hepatitis B (HBV), Hepatitis C (HCV), and Human Immunodeficiency Virus (HIV).
4. Have a negative urine hCG test if female of childbearing potential.
5. Able to swallow antibiotic, FMT or placebo capsules.
6. Able to give informed consent and/or assent as appropriate (patients 12-17 will be asked to provide written assent, patients 5-11 will be observed for assent or dissent behaviorally, or with verbal/written communication)
7. Willing and able to participate in the study requirements, including serial stool collection, survey completion and clinic visits.
8. Willing to undergo telephone follow-up to assess for safety and adverse events.
9. Must be free of any known food allergy.
10. Agrees and willing to have an enema for purposes of induction therapy.

Patients who have disease that has required other medications (including steroids, immunosuppressives, and biologics) will be included.

Exclusion Criteria:

Subjects who fall into any of the following exclusion criteria at the time of screening are not eligible for enrollment into the study.

1. Patients with extensive and/or severe CD (i.e. fistulizing disease, abscess, small bowel obstruction, fevers).
2. Patients in a clinical remission (PUCAI < 9) or (PCDAI <10).
3. Patients with recent (within 4 weeks) dose change of biologics, 5-ASA, steroids or immunomodulators
4. Patients considered to have toxic megacolon.
5. Patients with a known drug allergy to vancomycin, metronidazole or polymyxin.
6. Patients with a history of aspiration, gastroparesis, surgery involving the upper gastrointestinal tract (that might affect upper gastrointestinal motility) or unable to swallow pills.
7. Patients with esophageal dysmotility or swallowing dysfunction.
8. Patients with known food allergies.
9. Patients with positive test results for HBV, HCV, or HIV.
10. Female patients with a positive test result on a urine hCG test.
11. Patients unwilling or unable to give consent or participate in all study requirements.
12. Patients unable or unwilling to receive a retention enema for purposes of induction therapy.
13. Patients with recent (within 6 weeks) systemic antibiotic use.
14. Patients who have testing consistent with active clostridium difficile.
15. Patients with known prior experience with donor FMT.

Ages: 5 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 15 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2019-04-08 (Actual); Study Completion 2019-04-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stacy A Kahn, MD, Principal Investigator — Boston Childrens Hospital - GI & Nutrition
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Fecal Microbiota Transplant (FMT) | Placebo
Started | 10 | 5
Completed | 7 | 4
Not Completed | 3 | 1

BASELINE CHARACTERISTICS:
Population: There were two participants that were removed from the study after providing informed consent but before receiving any treatment. As a result, these participants were not included in the analysis and were not followed for adverse events.
Groups:
- Total: Total of all reporting groups
Arm/Group | Fecal Microbiota Transplant (FMT) | Placebo | Total
Number analyzed (Participants) | 8 | 5 | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 2 | 2 | 4
  Between 18 and 65 years | 6 | 3 | 9
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1
  Male | 8 | 4 | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 8 | 5 | 13
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 8 | 5 | 13

OUTCOME MEASURES:

1. Primary Outcome: 1. Safety and Tolerability of Universal Donor FMT Compared to Placebo: FMT-related Adverse Events Grade 2 or Above
Description: Number of participants with FMT-related adverse events grade 2 or above experienced in each arm.
Time Frame: At 8 weeks after start of FMT up to 6 months post treatment, an average of 10 months
Population: Participants who received FMT or placebo, completed the study, and follow up data is available.
Measure: Count of Participants; unit: Participants
Arm/Group | Fecal Microbiota Transplant (FMT) | Placebo
Number analyzed (Participants) | 8 | 5
Participants | 4 | 0

2. Secondary Outcome: Remission of Disease
Description: Remission as defined by a PUCAI score of less than 9 (for UC) or by a PCDAI score of less than 10 (for CD)
Time Frame: At all intermediate timepoints until 6 month follow up post intervention, an average of 10 months
Population: Participants who received FMT or placebo, completed the study, and follow up data is available.
Measure: Count of Participants; unit: Participants
Groups:
- Fecal Microbiota Transplant (FMT) Crohn's Disease: Participants with a diagnosis of Crohn's Disease that received induction retention enema for the first week of treatment followed by once weekly administration of 15 capsules of study treatment (the equivalent of 7.5 grams of human stool) will be (administered within 60 minutes of thawing once weekly) for 7 weeks. After completing 8 weeks of blinded study treatment, study subjects on FMT who have shown improvement will be given the option to receive open-label maintenance FMT weekly for an additional 8 weeks of once weekly FMT capsule administration.
  Fecal Microbiota Transplant (FMT): The study intervention consists of frozen, bottled or encapsulated fecal microbiota preparations that have been screened and prepared to a uniform and rigorous standard by OpenBiome. FMT is performed by patients receiving a retention enema and swallowing capsules, introducing stool from a healthy donor into their intestinal tract.
- Placebo Crohn's Disease: Participants with a diagnosis of Crohn's Disease that received induction placebo enema for the first week of treatment followed by once weekly administration of 15 capsules of study placebo (administered within 60 minutes of thawing once weekly) for 7 weeks. After completing 8 weeks of blinded study placebo, study subjects on placebo who DO NOT demonstrate improvement will be given the option to receive open-label maintenance FMT weekly for an additional 8 weeks, beginning with a FMT induction enema followed by 7 weeks of weekly FMT capsule administration.
  Placebo: Placebo administration will consist of both a placebo retention enema and placebo capsules.
- Fecal Microbiota Transplant (FMT) Ulcerative Colitis: Participants with a diagnosis of Ulcerative Colitis that received induction retention enema for the first week of treatment followed by once weekly administration of 15 capsules of study treatment (the equivalent of 7.5 grams of human stool) will be (administered within 60 minutes of thawing once weekly) for 7 weeks. After completing 8 weeks of blinded study treatment, study subjects on FMT who have shown improvement will be given the option to receive open-label maintenance FMT weekly for an additional 8 weeks of once weekly FMT capsule administration.
- Placebo Ulcerative Colitis: Participants with a diagnosis of Ulcerative Colitis that received induction placebo enema for the first week of treatment followed by once weekly administration of 15 capsules of study placebo (administered within 60 minutes of thawing once weekly) for 7 weeks. After completing 8 weeks of blinded study placebo, study subjects on placebo who DO NOT demonstrate improvement will be given the option to receive open-label maintenance FMT weekly for an additional 8 weeks, beginning with a FMT induction enema followed by 7 weeks of weekly FMT capsule administration.
Arm/Group | Fecal Microbiota Transplant (FMT) Crohn's Disease | Placebo Crohn's Disease | Fecal Microbiota Transplant (FMT) Ulcerative Colitis | Placebo Ulcerative Colitis
Number analyzed (Participants) | 1 | 2 | 5 | 3
Participants | 1 | 0 | 2 | 0

3. Secondary Outcome: Improvement in Inflammatory Biomarkers
Description: Improvement in inflammatory biomarkers (stool calprotectin, serum ESR, CRP, albumin, hematocrit) compared to baseline.
Time Frame: At End of Treatment (8 weeks) and at 6 month post treatment
Population: Participants who received FMT or placebo, completed the study, and follow up data is available.
Measure: Count of Participants; unit: Participants
Groups:
- Fecal Microbiota Transplant (FMT) at 8 Weeks After Treatment; Placebo Group After Open Label FMT: Induction retention enema for the first week of treatment followed by once weekly administration of 15 capsules of study treatment (the equivalent of 7.5 grams of human stool) will be (administered within 60 minutes of thawing once weekly) for 7 weeks. After completing 8 weeks of blinded study treatment, study subjects on FMT who have shown improvement will be given the option to receive open-label maintenance FMT weekly for an additional 8 weeks of once weekly FMT capsule administration.
  Fecal Microbiota Transplant (FMT): The study intervention consists of frozen, bottled or encapsulated fecal microbiota preparations that have been screened and prepared to a uniform and rigorous standard by OpenBiome. FMT is performed by patients receiving a retention enema and swallowing capsules, introducing stool from a healthy donor into their intestinal tract.
- Placebo at End of Treatment Before Open-Label FMT: Induction placebo enema for the first week of treatment followed by once weekly administration of 15 capsules of study placebo (administered within 60 minutes of thawing once weekly) for 7 weeks. After completing 8 weeks of blinded study placebo, study subjects on placebo who DO NOT demonstrate improvement will be given the option to receive open-label maintenance FMT weekly for an additional 8 weeks, beginning with a FMT induction enema followed by 7 weeks of weekly FMT capsule administration.
  Placebo: Placebo administration will consist of both a placebo retention enema and placebo capsules.
Arm/Group | Fecal Microbiota Transplant (FMT) at 8 Weeks After Treatment | Placebo at End of Treatment Before Open-Label FMT | Placebo Group After Open Label FMT
Number analyzed (Participants) | 6 | 5 | 4
Participants
  Decrease in Fecal Calprotectin at 8 weeks | 1 | 3 | 1
  Decrease in Fecal Calprotectin at 6 months | 1 | 0 | 2
  Decrease in CRP at 8 weeks | 1 | 2 | 0
  Decrease in CRP at 6 months | 1 | 0 | 1
  Decrease in ESR at 8 weeks | 0 | 0 | 0
  Decrease in ESR at 6 months | 2 | 0 | 0

4. Secondary Outcome: Percentage of Donor Microbiome Present in Transplant Recipient
Description: We will assess changes in microbial composition and the extent of microbial engraftment from the donor in the recipient by comparing the similarity of the microbiomes at two weeks at seven weeks after the induction enema.
Time Frame: At two weeks and seven weeks post induction enema
Population: Participants who received FMT or placebo, completed the study, and follow up data is available.
Measure: Mean (Full Range); unit: percentage of donor microbiome present
Groups:
- Open Label After Placebo: Open-Label treatment for those previously assigned to Placebo Group. Open-Label treatment included an induction retention enema for the first week of treatment followed by once weekly FMT capsules
Arm/Group | Fecal Microbiota Transplant (FMT) | Open Label After Placebo
Number analyzed (Participants) | 6 | 4
percentage of donor microbiome present
  Engraftment at 2 weeks | 74.8 [33.3 to 90.1] | 41.8 [26.2 to 64.9]
  Engraftment at 7 weeks | 68.3 [7.34 to 91.5] | 47.9 [2.8 to 84.4]

5. Secondary Outcome: Number of Participants With Improvement in Disease Activity
Description: 5a. For UC - Improvement of Pediatric Ulcerative Colitis Activity Index (PUCAI) by 20 points or more.
  Improvement in disease status as measured by improvement of PUCAI score by 20 points or more.
  5b. For CD - Improvement of Pediatric Crohn's Disease Activity Index (PCDAI) by 12.5 points or more.
  Improvement of disease status as measured by improvement of PCDAI score by 12.5 points or more.
Time Frame: At 8 weeks after start of FMT
Population: There were 1 CD and 5 UC participants in the FMT group that completed the study protocol and follow up. There were 2 CD and 3 UC participants that completed the Placebo and were eligible for 8 weeks of Open-Label FMT that completed the study protocol and follow up.
Measure: Count of Participants; unit: Participants
Groups:
- FMT After Placebo: Induction placebo enema for the first week of treatment followed by once weekly administration of 15 capsules of study placebo (administered within 60 minutes of thawing once weekly) for 7 weeks. After completing 8 weeks of blinded study placebo, study subjects on placebo who DO NOT demonstrate improvement will be given the option to receive open-label maintenance FMT weekly for an additional 8 weeks, beginning with a FMT induction enema followed by 7 weeks of weekly FMT capsule administration.
  Placebo: Placebo administration will consist of both a placebo retention enema and placebo capsules.
Arm/Group | Fecal Microbiota Transplant (FMT) | FMT After Placebo
Number analyzed (Participants) | 6 | 5
Participants
  UC Participants with improved disease scores as defined in outcome measure description: number analyzed (Participants) | 5 | 3
  UC Participants with improved disease scores as defined in outcome measure description | 2 | 0
  CD Participants with improved disease scores as defined in outcome measure description: number analyzed (Participants) | 1 | 2
  CD Participants with improved disease scores as defined in outcome measure description | 1 | 0
  UC and CD participants that did not meet improved disease activity score definitions | 3 | 5

ADVERSE EVENTS:
Time Frame: The adverse event data was collected for 1 year post treatment, up to approximately 1 year and 4 months.
Description: The definitions do not differ.
Groups:
- Fecal Microbiota Transplant (FMT): Adverse events are reported for participants during and after receiving FMT in either blinded or open-label treatment.
  Induction retention enema for the first week of treatment followed by once weekly administration of 15 capsules of study treatment (the equivalent of 7.5 grams of human stool) will be (administered within 60 minutes of thawing once weekly) for 7 weeks. After completing 8 weeks of blinded study treatment, study subjects on FMT who have shown improvement will be given the option to receive open-label maintenance FMT weekly for an additional 8 weeks of once weekly FMT capsule administration.
  Fecal Microbiota Transplant (FMT): The study intervention consists of frozen, bottled or encapsulated fecal microbiota preparations that have been screened and prepared to a uniform and rigorous standard by OpenBiome. FMT is performed by patients receiving a retention enema and swallowing capsules, introducing stool from a healthy donor into their intestinal tract.
- Placebo: Adverse events are reported for participants during receipt of placebo treatment.
  Induction placebo enema for the first week of treatment followed by once weekly administration of 15 capsules of study placebo (administered within 60 minutes of thawing once weekly) for 7 weeks. After completing 8 weeks of blinded study placebo, study subjects on placebo who DO NOT demonstrate improvement will be given the option to receive open-label maintenance FMT weekly for an additional 8 weeks, beginning with a FMT induction enema followed by 7 weeks of weekly FMT capsule administration.
  Placebo: Placebo administration will consist of both a placebo retention enema and placebo capsules.
Arm/Group | Fecal Microbiota Transplant (FMT) | Placebo
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/5
Serious Adverse Events (participants affected / at risk) | 3/12 | 0/5
Other Adverse Events (participants affected / at risk) | 6/12 | 1/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fecal Microbiota Transplant (FMT) (N=12) | Placebo (N=5)
Grade 3 Sinus Tachycardia (Cardiac disorders) | 1 (1) | 0 (0) — Hypersensitivity reaction from FMT induction enema resulting in sinus tachycardia and an ED admission. Inpatient for 2 days following
Grade 3 Colitis (Gastrointestinal disorders) | 2 (2) | 0 (0) — Increase in symptoms like abdominal pain, blood in stool and or watery stool, high frequency of stooling, nausea/vomiting, and dehydration
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fecal Microbiota Transplant (FMT) (N=12) | Placebo (N=5)
Epiploic Appendagitis (Gastrointestinal disorders) | 1 (1) | 0 (0) — AE was not related to study intervention.
Abnormal Lab Values (Immune system disorders) | 2 (12) | 0 (0) — Decreased WBC, increased bilirubin, increase Alkaline phosphatase, and increased lymphocyte count were all present but were determined to be not related or present at baseline.
Fever (General disorders) | 1 (1) | 1 (1) — Fever, dizziness, flushing, and chills were reported as probably related and resolved without sequelae
Eczema/Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) — Eczema and rash unrelated to the study treatment were reported
Sore Throat (Respiratory, thoracic and mediastinal disorders) | 1 (3) | 0 (0) — Sore Throat
Non-Cardiac Chest Pain (General disorders) | 2 (3) | 0 (0) — Non-Cardiac Chest Pain
Upper Respiratory Infection (Respiratory, thoracic and mediastinal disorders) | 1 (3) | 0 (0) — Upper Respiratory Infection
Eye Disorder/Blurred Vision (Eye disorders) | 1 (2) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-05-11): https://cdn.clinicaltrials.gov/large-docs/53/NCT02330653/Prot_SAP_000.pdf